CLINICAL TRIAL: NCT05424510
Title: Prevention of Hypotension After Induction of General Anesthesia Using POint-of-care Ultrasound to Guide Fluid Management: a Randomized Controlled Trial
Brief Title: PoCUS Guided Fluids to Prevent Post-induction Hypotension
Acronym: HIPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, James Khan, Pain Physician and Anesthesiologist, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 22-0043-A
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Hypotension on Induction
Keywords: point of care ultrasound; general anesthesia
MeSH Terms: interventions — Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: Based on the IVC PoCUS exam, volume responsive patients will be randomized into two equal groups: half will receive a fluid bolus (FB+) and half will not (FB-). Patients in the FB+ group will receive a single bolus of 500 ml of Ringer's Lactate over 5-10 minutes with an additional IVC scan at the end of the infusion to record the change in IVC-CI.
Who Masked: Care Provider
Masking Description: In all fluid responsive patients an IV line will be placed, regardless of group allocation into FB+ or FB-. In order to maintain masking of the treating anesthesiologist, patients will be advised regarding the importance to not disclose whether they received a fluid bolus or not to their anesthetist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluid Bolus (FB+) (Active Comparator): Patients in the FB+ group will receive a single bolus of 500 ml of Ringer's Lactate over 5-10 minutes.
  Interventions: Drug: Ringer's Lactate; Other: IV line
- Non fluid bolus (FB-) (Placebo Comparator): Patients in the FB- group will not receive a fluid bolus.
  Interventions: Other: IV line

INTERVENTIONS:
Drug: Ringer's Lactate — 500 ml of Ringer's Lactate
  Arms: Fluid Bolus (FB+)
Other: IV line — Placing of an IV line before surgery

SUMMARY:
Hypotension is a common side-effect of general anesthesia induction, and is related to adverse outcomes, including a significantly increased risk of one-year mortality. Hypovolemia is a significant risk factor, and optimized fluid therapy remains the cornerstone of its treatment. Ultrasound measurements of inferior vena cava (IVC) diameter with respiration have been recommended as rapid and noninvasive methods for estimating volume status. Several recent studies reported that preoperative IVC ultrasound has a reliable predicting ability of arterial hypotension after the induction of general anesthesia. The practical effect of optimizing fluid status before surgery using this ability has not been studied. Our hypothesis is that preoperative ultrasound-guided intravenous fluid bolus administration may reduce the incidence of hypotension after the induction of general anesthesia in adults presenting for elective non-cardiac, non-obstetric surgery

DETAILED DESCRIPTION:
Background: Hypotension is a common side-effect of general anesthesia induction, and is related to adverse outcomes, including significantly increasing risk of one-year mortality (intraoperative systolic hypotension increased mortality risk by 3.6% per minute below 80 mm Hg). Even short durations of intraoperative hypotension have been associated with acute kidney injury (AKI) and myocardial injury.

The feasibility of POCUS in directing fluid management to prevent hypotension has been demonstrated after the induction of spinal anesthesia but not general anesthesia.

Design: This will be a randomized controlled trial. All participating patients will undergo a bed-side ultrasound scan and assessment of the IVC-CI. Patients with collapsible IVC, defined as a CI equal or greater than 43%, will be randomized 1:1 to either receive a fluid bolus or not. We will test the potential efficacy of an ultrasound directed fluid bolus in reducing the hypotension associated with the induction of general anesthesia. This will be a single blinded study with the attending anesthesiologist unaware to patient group allocation and POCUS data.

The primary objective is to determine the efficacy of preoperative POCUS-guided intravenous fluid bolus administration in reducing the incidence of hypotension after the induction of general anesthesia in adults presenting for elective non-cardiac, non-obstetric surgery.

While in the preoperative area, patients who fulfil the eligibility criteria will be approached for recruitment, informed consent, and voluntary participation. Written informed consent will be obtained from all patients. Upon informed consent, baseline characteristics will be collected which include demographic information, past medical history including medical therapy, and the type of scheduled surgery. Thereafter the assessment of preoperative IVC-CI will be performed, with patients with an IVC-CI ≥ 43% randomized into the intervention and control groups.

Randomization: Patients who fulfil the eligibility criteria, provide informed consent, and are found to have an IVC-CI ≥ 43% according to a POCUS assessment, will be randomized prior to surgery while in the preoperative area. The allocation sequence will be created by a statistician through a computer-generated random table, and concealed in sequentially numbered, opaque, sealed envelopes, with a 1:1 allocation ratio and random block sizes of 4, 6, and 8 participants. Attending clinicians involved in the care of the patient will be blinded to the allocation and intervention.

Data collected in the preoperative area will include patient demographics [gender, age, height, weight, past medical history including coronary artery disease, heart failure, diabetes, smoking, peripheral vascular disease, hypertension, current treatment with beta-blockers, ACE-I or ARBs, and diuretics, type of surgery (coded as lower limb or upper limb orthopedic surgery, lower abdominal surgery, vascular, gynecology (non-obstetric) and urology), and the preoperative fasting duration.

In addition to the IVC measurements obtained by the POCUS scan, we will also document the duration of the POCUS scan and the fluid bolus administration, as well as the baseline perfusion index (PI), which estimates the pulsatility of blood in the extremities, calculated using infrared spectrum as part of plethysmography waveform processing, and has been shown to predict hypotension following propofol induction.

Once in the operating room, the information from the induction of the general anesthesia will be collected through the routine electronic chart including blood pressure and heart rate (before the induction of anesthesia), drugs administered during and after induction, and blood pressure over 20 minutes from the start of induction. In case of an arterial line inserted before induction to measure blood pressure invasively and continuously, which is indicated according to the discretion of the treating anesthesiologist, it will be used to collect the blood pressure and heart rate information.

A previously reported IVC-CI threshold of 43% had a positive predicting value (PPV) of 86% in predicting post-induction hypotension. As our sample will only include patients with a collapsible IVC (IVC-CI ≥ 43%), for the sample size calculation we will assume a 85% incidence of post-induction hypotension in the FB- group. Since no prior studies have assessed the effect of IVC-CI guided fluid bolus within the general anesthesia population, we will choose a relative risk reduction (RRR) of 50% with POCUS directed fluid optimization as clinically significant. Thus, assuming post-induction hypotension incidence of 85% and 42.5% in the FB- and FB+ groups, respectively, a sample size of 19 patients per group (95% confidence level) is required to reject the null-hypothesis with a risk of 0.05 and a power of 0.8.

Statistical analysis will follow the trial completion. No other interim analysis will occur during this trial. Data collected during the study will be compiled using Excel spreadsheets (Microsoft, USA). The lowest MAP recorded during the twenty minutes after the start of induction, defined as the first administration of an anesthetic agent at an anesthetic dosage, will be used to calculate the percentage decrease from baseline in each patient. Baseline will be defined as the first blood pressure measurement in the preoperative area or from the pre-anesthesia clinic visit. Descriptive data will be presented as means ± standard deviation (SD) for continuous variables and as absolute numbers and percentages for categorical variables. This data will include patient demographics, IVC-CI, the incidence of hypotension and its total duration, the total amount of fluids and vasopressors administered, the mean duration of the POCUS scan, and the incidence of surgical delays. For our primary outcome, the reduction in the incidence of post-induction hypotension between FB+ and FB- groups, we will use a χ2 test. Student's t test will be used for parametric data null hypothesis testing, while two-tailed Manne Whitney U test will be used to evaluate significance in non-normally distributed parameters.

In all cases a p value < 0.05 will be considered as statistically significant. Statistical analysis will be performed using SPSS version 20 (IBM, Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Elective surgery
* IVC-CI ≥ 43% on their preoperative POCUS scan.

Exclusion Criteria:

* Hypotension, defined as MAP below 65 mmhg, prior to the induction of general anesthesia.
* Treated with angiotensin converting enzyme inhibitors (ACE-I) or angiotensin receptor blockers (ARB) on the day of surgery.
* Patients with heart failure with ejection fraction (EF) < 40%.
* Patients with documented acute or chronic renal failure.
* Patients with neuraxial blockade (epidural or spinal) performed before induction of general anesthesia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
Difference in the incidence of hypotension after induction of general anesthesia | 20 minutes from the induction of general anesthesia
  hypotension as MAP below an absolute threshold of 65 mmhg or relative threshold of 25% decrease from baseline, or the administration of vasopressors during the induction period

SECONDARY OUTCOMES:
The incidence of surgical delays | Patient consent until the beginning of the operation
  any occurrence where the treating surgical or anesthetic team asked to transfer the patient to the OR but were subject to delay stemming from the POCUS assessment or the fluid bolus
The duration of post-induction hypotension | 20 minutes after induction
  The duration of from the first hypotension measurement recorded until it was resolved. In case there are several occurrences of hypotension during this period, its total duration will be summed.
Adverse events | 20 minutes after induction
  Adverse events such as pulmonary edema recorded throughout the induction period.

CONTACTS AND LOCATIONS:
Overall Officials: James S Khan, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dana E, Arzola C, Khan JS. Prevention of hypotension after induction of general anesthesia using point-of-care ultrasound to guide fluid management: a randomized controlled trial. Can J Anaesth. 2024 Sep;71(9):1219-1228. doi: 10.1007/s12630-024-02748-8. Epub 2024 Mar 13. PMID 38480632